CLINICAL TRIAL: NCT00615095
Title: Differential Risks for Melanoma: p16 and DNA Repair
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of New Mexico (Other); Yale University (Other)
Responsible Party: IRENE ORLOW, PH.D., M.S., Memorial Sloan-Kettering Cancer Center
Other Study IDs: 97-012
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Melanoma; Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (3):
- 1: Cases will be patients 18 years or older with a histologically confirmed, second or multiple primary melanoma.
  Interventions: Other: self-administered questionnaire and blood draw
- 2: Controls will be patients 18 years or older with a histologically confirmed first primary melanoma diagnosed no earlier than 12 months prior to the study start date.
  Interventions: Other: self-administered questionnaire and blood draw
- 3: Healthy controls will be subjects 18 years or older recruited from the general population through random digit dialing. These subjects will have no history of melanoma. They will also be frequency matched to cases on the basis of sex and 10-year age group.
  Interventions: Other: health questionnaire, blood draw and skin exam

INTERVENTIONS:
Other: self-administered questionnaire and blood draw — Epidemiologic data will be collected via a self-administered questionnaire which will be distributed to subjects by a member of the study staff. It should take less than fifteen minutes to complete, and subjects will have the options of completing it at the time of their blood-drawing or filling it out at home and mailing it back to the study staff.
  Groups: 1
Other: self-administered questionnaire and blood draw — Epidemiologic data will be collected via a self-administered questionnaire which will be distributed to subjects by a member of the study staff. It should take less than fifteen minutes to complete, and subjects will have the options of completing it at the time of their blood-drawing or filling it out at home and mailing it back to the study staff.
  Groups: 2
Other: health questionnaire, blood draw and skin exam — Numbers will be randomly selected from a pool of prefixes. Numbers will be screened by computer for being working, non-business, non-fax, and non-modem numbers. After establishing eligibility for the study, we will send the potential control a letter further explaining the purpose of the study and its requirements. An interviewer will then call to arrange an appointment. During the interview, the subject will sign informed consent, be given the public health questionnaire, have 30 ml of blood drawn, and undergo the skin examination of arms and back.
  Groups: 3

SUMMARY:
The goal of this study is to find out if some people are more likely to get melanoma, a form of skin cancer, than others. People respond to the environment in different ways. Some may be born with genes that make them more likely to get this type of skin cancer. Genes are made up of DNA. DNA damage is one of the first steps in developing cancer. Each person has many ways to repair normal damage to their genes. Some people may have a lower level of this repair and that may make them more likely to get cancer. Some genes are important for DNA repair. The genes we want to test are thought to affect the rate at which DNA can be repaired. We also want to find out if sun habits are related to these levels of DNA repair or genetic mutations.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be patients 18 years or older with a histologically confirmed, second or multiple primary melanoma. These will be sequentially selected from subjects seen at Memorial Sloan-Kettering Cancer Center or the Yale University Pigmented Lesion Clinic.
* Controls will be patients 18 years or older with a histologically confirmed first primary melanoma diagnosed no earlier than 12 months prior to the study start date. One control will be selected per case. These patients will be referred to the study by the Melanoma Disease Management Team at Memorial Sloan-Kettering Cancer Center. Controls will be frequency-matched to cases on the basis of sex and age (within 10 year age groups).
* Healthy controls will be subjects 18 years or older recruited from the general population through random digit dialing. These subjects will have no history of melanoma. They will also be frequency matched to cases on the basis of sex and 10-year age group.
* The subject must have a histologically confirmed malignant melanoma.
* Cases may have an in situ melanoma as the second primary.
* Melanoma Controls may have only one primary melanoma.
* Healthy controls should have no history of melanoma.
* The subject's physician consents to his/her patient's participation in the study (if the subject has a diagnosis of melanoma).
* The subject has consented, in writing, to participate in the study

Exclusion Criteria:

* Karnofsky status less than 60 (see Appendix). This will be evaluated by the physician treating the subject for melanoma at the time permission is given for participation
* Patient had chemotherapy or radiation therapy within the last 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Second or multiple primary melanoma cases will be identified at Memorial Sloan-Kettering Cancer Center, the Yale University Pigmented Lesion Clinic, or from among those subjects who participated in the earlier case-control study in Connecticut.
  First primary melanoma cases will be identified and referred to the study staff by participating physicians on the Melanoma Disease Management Team at Memorial Sloan-Kettering Cancer Center.
  Random digit dialing will be used to locate 100 population-based controls for this study. We will use telephone prefixes in Connecticut
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 1997-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
evaluate the relative risks of develop melanoma for those individuals with deficient DNA repair in a case-control study of multiple primary melanoma, where the controls are cases of first primary melanoma & healthy subjects from the general population. | conclusion of study

SECONDARY OUTCOMES:
is to investigate associations of specific polymorphisms of the melanocortin receptor gene with clinical cutaneous phenotype (hair color, eye color, skin color, and freckling tendency). | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Irlene Orlow, PH.D., M.S., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org